CLINICAL TRIAL: NCT04679298
Title: Qualitative Coagulation Testing With the CoaguChek(R) Pro II Point-of-Care Test System and aPTT Test Cards in Patients Before and After First Intake of Direct Oral Anticoagulants
Brief Title: Point-of-Care Testing of Coagulation in Patients Treated With Direct Oral Anticoagulants Extended
Acronym: POCT-DOAC ext
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Heart and Diabetes Center North Rhine-Westphalia (Other)
Responsible Party: Sponsor
Other Study IDs: 703/2020BO1
Record Dates: First submitted 2020-12-16; First posted 2020-12-22 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Anticoagulation With Direct Oral Anticoagulants
Keywords: Direct oral anticoagulants; Acute stroke; Point-of-care testing
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Apixaban: N=20
- Edoxaban: N=20
- Dabigatran: N=20
- Rivaroxaban: N=20

SUMMARY:
The investigators' study aims to test the correlation between CoaguChek point-of-care aPTT testing (Roche, Switzerland) and low plasma levels of all four currently EMA approved direct oral anticoagulants (DOAC; apixaban, dabigatran, edoxaban, and rivaroxaban) and to determine the diagnostic accuracy of POCT to rule out or detect relevant levels of DOAC in real-life stroke patients. Relevant levels are defined as current treatment thresholds according to international guidelines, i.e. 30 and 50 ng/mL.

DETAILED DESCRIPTION:
In emergency situations such as an acute stroke or emergency surgery, information on the plasma concentration of DOAC in patients with suspected or known intake of DOAC plays a vital role in making decisions in relation to the administration of i.v thrombolysis therapy- ''Time is brain'' or to consider the administration of an antidote in acute hemorrhagic stroke patients. Moreover, acute stroke patients presenting with aphasia are not in the position to provide information on how regular and when last the anticoagulant was taken.

Although dabigatran for example has lab tests such as the diluted thrombin time (dTT) and the ecarin clotting time (ECT) available, major challenges faced are due to the scarcity of these tests in many hospitals. Also, just like many other lab tests, results could take up to 30-60 minutes (turn-around time due to transport and sample processing) making it inconvenient in critical situations.

In our previous studies, we have been able to show a concentration-dependent effect of Dabigatran on Hemochron® Signature POCT (Werfen, Barcelona, Spain) with all 4 test cards used (PT, aPTT, ACT-LR und ACT+). Dabigatran however failed to show a concentration-dependent effect when tested with the CoaguChek®XS Pro POCT device (Roche, Switzerland) together with the then available prothrombin time (PT) test card. This finding could be attributed to the known low response of dabigatran plasma levels on PT but rather a better response of dabigatran plasma levels on aPTT.

Our study therefore aims to test CoaguChek® Pro II POCT device which is widely available in Europe with the new aPTT test card on all 4 DOAC in order to assess a possible correlation between the aPTT values and the DOAC plasma concentration detected by mass spectrometry, and to evaluate its ability to rule out even very low but clinically relevant DOAC concentrations (e.g., above the currently recommended 30 and 50 ng/mL treatment thresholds). In order to avoid POCT results indicating no relevant DOAC concentrations despite DOAC concentrations being actually elevated, our specificity target is predefined as >95% for detection of elevated DOAC concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Stroke patients, who were newly started on oral anticoagulation with apixaban, edoxaban, dabigatran or rivaroxaban for secondary prevention of thromboembolic events
* informed consent

Exclusion Criteria:

* Vitamin K antagonists ≤ 14 days prior to study participation
* Prior DOAC intake ≤ 72 hours
* Low-molecular weight heparin ≤ 24 hours
* Unfractionated heparin ≤ 12 hours
* Heparinoids (e.g. Fondaparinux) ≤ 72 hours
* Abnormal coagulation values at baseline (Quick < 70% or activated thromboplastin time (aPTT) > 40sec.)
* History of coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive stroke patients, who were newly started on oral anticoagulation with apixaban, edoxaban, dabigatran or rivaroxaban for secondary prevention of thromboembolic events
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Effect/Correlation of direct oral anticoagulants (DOAC) on aPTT CoaguChek® Pro II point-of-care testing (POCT) result | 24 hours
  DOAC concentrations will be determined by ultra-performance liquid chromatography-tandem mass spectrometry

SECONDARY OUTCOMES:
Diagnostic accuracy of the CoaguChek® Pro II POCT to rule out or detect relevant DOAC levels | 24 hours
  aPTT test card specificity and sensitivity do rule out or detect relevant DOAC plasma concentrations
Effect/Correlation of DOAC on calibrated DOAC-specific coagulation assays | 24 hours
  Response of calibrated anti-thrombin/Xa activity assays to dabigatran/factor Xa inhibitors' plasma levels

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

REFERENCES:
- [Background] Ebner M, Birschmann I, Peter A, Hartig F, Spencer C, Kuhn J, Blumenstock G, Zuern CS, Ziemann U, Poli S. Emergency Coagulation Assessment During Treatment With Direct Oral Anticoagulants: Limitations and Solutions. Stroke. 2017 Sep;48(9):2457-2463. doi: 10.1161/STROKEAHA.117.017981. Epub 2017 Aug 3. PMID 28775134
- [Background] Ebner M, Birschmann I, Peter A, Spencer C, Hartig F, Kuhn J, Blumenstock G, Zuern CS, Ziemann U, Poli S. Point-of-care testing for emergency assessment of coagulation in patients treated with direct oral anticoagulants. Crit Care. 2017 Feb 15;21(1):32. doi: 10.1186/s13054-017-1619-z. PMID 28196509
- [Background] Ebner M, Peter A, Spencer C, Hartig F, Birschmann I, Kuhn J, Wolf M, Winter N, Russo F, Zuern CS, Blumenstock G, Ziemann U, Poli S. Point-of-Care Testing of Coagulation in Patients Treated With Non-Vitamin K Antagonist Oral Anticoagulants. Stroke. 2015 Oct;46(10):2741-7. doi: 10.1161/STROKEAHA.115.010148. Epub 2015 Aug 13. PMID 26272385
- [Background] Hartig F, Birschmann I, Peter A, Horber S, Ebner M, Sonnleitner M, Spencer C, Bombach P, Stefanou MI, Kuhn J, Mengel A, Ziemann U, Poli S. Point-of-care testing of coagulation in patients treated with edoxaban. J Thromb Thrombolysis. 2020 Oct;50(3):632-639. doi: 10.1007/s11239-020-02143-2. PMID 32436010